CLINICAL TRIAL: NCT00566085
Title: Molecular Breast Imaging: Evaluation of a New Technique Using Scintimammography as an Additional Diagnostic Tool for Women Undergoing Neoadjuvant Therapy for Breast Cancer - A Pilot Study
Brief Title: New Technique as an Additional Diagnostic Tool for Women Undergoing Neoadjuvant Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-002067
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: MBI; Breast Cancer; Neoadjuvant Therapy; Molecular Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Molecular Breast Imaging (Other)
  Interventions: Procedure: Molecular Breast Imaging

INTERVENTIONS:
Procedure: Molecular Breast Imaging — A dual-detector cadmium-zinc-telluride gamma camera system mounted on a modified mammography gantry is used to image the breast. The injection dose of the radiopharmaceutical given to the patient is 28-32 mCi of 99m Tc-sestamibi.
  Other Names: MBI

SUMMARY:
Molecular Breast Imaging is a highly promising novel methodology for breast cancer detection. Preliminary patient studies with our dual-detector system indicate that this system is capable of reliably detecting very small (5-10 mm) malignant lesions in the breast. Besides the usefulness of Molecular Breast Imaging for tumor detection, we speculate that tumor uptake and washout may be predictors to response to neoadjuvant therapy for patients with the diagnosis of breast cancer. We propose that in patients with breast cancer who undergo neoadjuvant chemotherapy or neoadjuvant hormone therapy that molecular breast imaging is an accurate test for assessing response rate to neoadjuvant therapy.

DETAILED DESCRIPTION:
Adjuvant therapy after surgery for breast cancer has provided significant benefits to patients at risk for relapse. However, the success of therapy for each individual patient will often take years to reveal. Preoperative (neoadjuvant) medical therapy is very potent as an initial treatment for inoperable and large operable breast cancers. Tumor regression can be achieved in the great majority of patients and downstaging frequently reduces the need for mastectomy and it has become clear that pathologic complete response is a good prognostic marker. Data from current trials suggest that survival is at least as good with preoperative as with postoperative neoadjuvant therapies (1). With this observation preoperative medical therapy has the advantage over post-operative neoadjuvant therapy that it can be used as a short term surrogate marker for long-term outcome. With this translational approach, the therapy for each patient can be more targeted and individualized leading to higher success rates; and further, new therapies for early breast cancer can be assessed much more quickly than is currently possible through protracted trials of neoadjuvant therapy (2). This approach is therefore being increasingly utilized in patients with lower stage breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 - 90
* Women with breast cancer scheduled to undergo neoadjuvant chemotherapy therapy or neoadjuvant hormone therapy
* Women who have undergone any breast imaging procedure, and in whom a repeat imaging procedure is planned prior to definite surgery

Exclusion Criteria:

* Pregnant or lactating
* Unable to understand or sign a consent form
* Physically unable to sit upright and still for 40 minutes

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To document that pre- and post-neoadjuvant therapy tumor size can be satisfactorily assessed by molecular breast imaging and corresponds to tumor size evaluation by conventional breast imaging procedures (mammogram, ultrasound, MRI). | Up to 6 months

SECONDARY OUTCOMES:
To document that post-neoadjuvant tumor size as determined by molecular breast imaging corresponds to tumor size found at time of surgery. | Up to 6 months
To characterize patterns of tumor uptake and washout and determine if they are predictors of response to neoadjuvant chemotherapy or neoadjuvant hormone therapy. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Smith IE, Lipton L. Preoperative/neoadjuvant medical therapy for early breast cancer. Lancet Oncol. 2001 Sep;2(9):561-70. doi: 10.1016/S1470-2045(01)00490-9. PMID 11905711
- [Background] Chow LW, Yiu CC, Yip AY, Loo WT. The future perspectives of breast cancer therapy. Biomed Pharmacother. 2006 Jul;60(6):259-62. doi: 10.1016/j.biopha.2006.06.010. Epub 2006 Jun 23. PMID 16824726